CLINICAL TRIAL: NCT00283036
Title: Efficacy and Tolerability of Posology Adaptation of Irbesartan in Ambulatory Hypertensive Patients
Brief Title: APROVE : Irbesartan in Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L_8793
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan

INTERVENTIONS:
Drug: Irbesartan

SUMMARY:
Study objective : To compare efficacy and tolerability of posology adaptation of Irbesartan in ambulatory Hypertensive patients

ELIGIBILITY:
Inclusion Criteria:

* Patient with mild or moderate hypertension defined with arterial diastolic pressure (PAD) at sit position between 90 mmHg and 110 mmHg and arterial systolic pressure (PAS) at sit position between 140 mmHg and 180 mmHg.
* Patient diagnosed after 3 consultations within 2 months who has never been under treatment and responding to the required conditions for hypertension treatment with irbesartan. This patient must has been under proper but insufficient hygieno dietetic diet
* Patient who has been under a none satisfied antihypertensive treatment, and for whom this treatment was stopped at least 2 weeks prior to inclusion.
* Patient with a laboratory analysis (urinary sediment- Na -K- creatinine, total cholesterol) and ECG during the month prior to inclusion.

Exclusion Criteria:

* Severe Hypertension defined by PAS > 180mmHg and/or PAD > 110 mmHg.
* Isolated systolic Hypertension
* Secondary Hypertension
* Arterial stenosis on unique kidney - arterial bilateral kidney stenosis
* Non-surgically sterilized women or non-menopaused women.
* Confirmed sodic depletion.
* Hypersensitivity to Irbesartan.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2005-04

PRIMARY OUTCOMES:
Arterial Tension
Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Nabil BENOUNICHE, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Algiers, Algeria